CLINICAL TRIAL: NCT06429722
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Pilot Study to Evaluate the Effects of Oral NMRA-335140 Versus Placebo in Participants With a Major Depressive Episode Associated With Bipolar II Disorder
Brief Title: To Evaluate the Effects of NMRA-335140 on Symptoms of Major Depression in Participants With Bipolar II Disorder.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neumora Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMRA-335140-202
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Episode Associated With Bipolar II Disorder
Keywords: NMRA-335140; Navacaprant; BTRX-335140; CYM-53093; Bipolar II Disorder; Major Depressive Episode; Placebo-controlled; Double-blind; NMRA335140; NMRA 335140
MeSH Terms: conditions — Bipolar Disorder | interventions — BTRX-335140

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor will also be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NMRA-335140 80 milligrams (mg) once daily (QD) (Experimental): Participants will receive a NMRA-335140 tablet at a dose of 80 mg QD.
  Interventions: Drug: NMRA-335140 80 mg
- Placebo (Placebo Comparator): Placebo participants will receive matching placebo tablet once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NMRA-335140 80 mg — Participants will receive NMRA-335140 at a dose of 80 mg QD, orally.
  Other Names: BTRX-335140; CYM-53093; Navacaprant
  Arms: NMRA-335140 80 milligrams (mg) once daily (QD)
Drug: Placebo — Placebo will be administered orally
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled pilot study aiming to evaluate the effects of NMRA-335140 on symptoms of major depression in adults with Bipolar (BP) II disorder. The study design consists of a Screening Period (up to 28 days), a 6-week Treatment Period (during which participants will receive either NMRA-335140 or placebo), and a 6-week Safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

1. Have a primary Diagnostic and Statistical Manual of Mental Disorders Fifth Edition Text Revised (DSM-5-TR) diagnosis of BP II disorder with a current major depressive episode (MDE), without psychotic features confirmed by Structured Clinical Interview for DSM 5 Disorders, Clinical Trials Version (SCID-5-CT) at screening (this may be a first or recurrent episode).
2. Participant's current MDE and lifetime history of hypomanic episodes must be confirmed by independent assessment.
3. The symptoms of the current MDE have been present for more than 4 weeks prior to the Screening Visit, but no longer than 12 months prior to the Screening Visit.
4. Have a MADRS total score of 25 or higher at Screening and Baseline.
5. A change in MADRS total score between Screening and Baseline of ≤20%.

Exclusion Criteria:

1. Have failed 2 or more courses of antidepressant (adequate dose and duration, i.e., minimum 6 weeks) or mood stabilizer/antipsychotic treatment (each or in combination) for treatment of depressive symptoms in the current MDE.
2. Have currently or in the past year any of the following DSM-5-TR disorders: bipolar episodes with mixed features (including the current MDE), bipolar II with rapid cycling pattern (4 or more distinct mood episodes during a 12-month period). Participants with comorbid generalized anxiety disorder, social anxiety disorder, simple phobias, panic disorder, for whom bipolar II MDE is considered the primary diagnosis are not excluded.
3. Have a lifetime diagnosis of bipolar I disorder (manic episode schizophrenia, schizoaffective disorder, schizophreniform disorder, anorexia nervosa, bulimia nervosa, cluster B personality disorder, post-traumatic stress disorder (PTSD), or obsessive- compulsive disorder.
4. Have moderate to severe substance or alcohol use disorder, per DSM-5-TR criteria, within the 12 months prior to screening (excluding nicotine).
5. Are actively suicidal (e.g., any suicide attempts within the past 12 months) or are at serious suicidal risk as indicated by any current suicidal intent, including a plan, as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) (score of "YES" on suicidal ideation Item 4 or 5 within 3 months prior to Visit 1 [screening]) and/or based on clinical evaluation by the Investigator; or are homicidal, in the opinion of the Investigator.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 6 in the Montgomery-Asberg Depression Rating Scale (MADRS) total score | Baseline and up to Week 6
  The MADRS is a 10-item, clinician-rated scale that evaluates the participant's depressive symptomatology during the past week. Participants are rated on items assessing feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each item will be scored on a 7- point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity. Thus, scores in the MADRS range from 0 to 60, with increasing scores indicating increasing severity.

SECONDARY OUTCOMES:
Change from Baseline to Week 6 assessed in the Snaith-Hamilton Pleasure Scale (SHAPS) total score | Baseline and up to Week 6
  The SHAPS is a 14-item participant-reported instrument which measures anhedonia. It has been shown to be valid and reliable in normal and clinical samples, with adequate construct validity, satisfactory test-retest reliability, and high internal consistency. The scale will be completed by the participant and reviewed by site personnel qualified to oversee completeness. Each of the 14 items has a set of 4 responses, 2 of which endorse agreement (Definitely Agree, Agree) and 2 of which endorse disagreement (Disagree, Strongly Disagree). A total score can be derived by summing the response items; where those answered with "strongly agree" will be coded as a 1, while a "strongly disagree" response will be coded as 4. Therefore, scores on the SHAPS can range from 14 to 56, with higher scores corresponding to higher levels of anhedonia.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Neumora Investigator Site, Phoenix, Arizona
  - Neumora Investigator Site, Little Rock, Arkansas
  - Neumora Investigator Site, Garden Grove, California
  - Neumora Investigator Site, Long Beach, California
  - Neumora Investigator Site, San Jose, California
  - Neumora Investigator Site, Torrance, California
  - Neumora Investigator Site, Gainesville, Florida
  - Neumora Investigator Site, Lauderhill, Florida
  - Neumora Investigator Site, Maitland, Florida
  - Neumora Investigator Site, Miami, Florida
  - Neumora Investigator Site, Miami Lakes, Florida
  - Neumora Investigator Site, Marietta, Georgia
  - Neumora Investigator Site, Savannah, Georgia
  - Neumora Investigator Site, Watertown, Massachusetts
  - Neumora Investigator Site, Flowood, Mississippi
  - Neumora Investigator Site, Marlton, New Jersey
  - Neumora Investigator Site, Princeton, New Jersey
  - Neumora Investigator Site, Toms River, New Jersey
  - Neumora Investigator Site, Brooklyn, New York
  - Neumora Investigator Site, Houston, Texas
  - Neumora Investigator Site, Bellevue, Washington